CLINICAL TRIAL: NCT04528862
Title: RESTART Trials: Reducing Error in ER Settings Through Attention Restoration Theory
Brief Title: Reducing Error in ER Settings Through Attention Restoration Theory
Acronym: RESTART
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to logistical issues the study as designed was determined to not be feasible.
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HM20019844
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Attention Fatigue, Attention Restoration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nature (Experimental)
  Interventions: Behavioral: Nature slides
- Urban (Sham Comparator)
  Interventions: Behavioral: Urban slides

INTERVENTIONS:
Behavioral: Nature slides — participants will view a presentation of nature slides
  Arms: Nature
Behavioral: Urban slides — participants will view a presentation of urban slides
  Arms: Urban

SUMMARY:
The purpose of this research study is to find out about how looking at different types of pictures can affect people's attention spans. Attention Restoration Theory (ART) suggests that there are two types of attention. One type (directed attention) can become tired and cause people to make mistakes. The other type (involuntary attention) gives directed attention a chance to rest, so people make less mistakes. Certain types of pictures are good at capturing involuntary attention. We think that capturing involuntary attention will help emergency physicians make less mistakes on tests of attention. This study will allow us to learn more about it.

DETAILED DESCRIPTION:
In this study, participants will be asked to do the following things:

1. Before their usual shift in the emergency department, arrive ten minutes early to rate their mood and complete a Digit Span Backwards (DSB) task that tests their memory of different sets of numbers.
2. Five hours into their shift, they will take a ten minute break.
3. During this break, they will be randomly assigned to view either a picture presentation of nature slides or urban slides.
4. After the presentation, they will complete the Digit Span Backwards task again, they will rate their mood again, then return to their shift.

Participation in this study will last up to 30 minutes. Approximately fifty individuals will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

• Emergency Medicine Resident of any PGY level. (1-5)

Exclusion Criteria:

* Anybody under the age of 18
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Working memory | 5 hours
  Working memory will be assessed using the Digit Span test. Participants are read a sequence of numbers and asked to repeat the same sequence back to the examiner in order (forward span) or in reverse order (backward span). Number of correctly repeated numbers is summed to yield a score ranging from 0 to 28. Higher scores indicated better working memory
Positive mood | 5 hours
  Positive mood will be assess using the positive affect (PA) scale of the Positive and Negative Affect Schedule (PANAS). The PA scale consists of 10 adjectives which are rated on a 5 point scale from slightly or not at all to extremely. Items are summed to yield a score ranging from 10 to 50 with higher number indicating higher affect.
Negative mood | 5 hours
  Negative mood will be assess using the negative affect (NA) scale of the PANAS. The NA scale consists of 10 adjectives which are rated on a 5 point scale from slightly or not at all to extremely. Items are summed to yield a score ranging from 10 to 50 with higher number indicating higher affect.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Miller, DO, Principal Investigator — Virginia Commonwealth University

IPD SHARING:
Plan to Share IPD: No